CLINICAL TRIAL: NCT05449171
Title: Efficacy of the Association of Hyaluronic Acid With High Molecular Weight, α-lipoic Acid (ALA), Magnesium, Vitamin B6 and Vitamin D, in the Prevention of Spontaneous Abortion in Patients at Risk
Brief Title: High Molecular Weight Hyaluronic Acid, α-lipoic Acid, Magnesium, Vitamin B6 and Vitamin D, in the Prevention of Spontaneous Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HA-PREV_22
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Abortion, Spontaneous
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Thioctic Acid; Magnesium; Vitamin B 6; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Treatment group (Experimental)
  Interventions: Other: high molecular weight hyaluronic acid, α-lipoic acid (ALA), magnesium, vitamin B6 and vitamin D

INTERVENTIONS:
Other: high molecular weight hyaluronic acid, α-lipoic acid (ALA), magnesium, vitamin B6 and vitamin D — Patients will take an association of high molecular weight hyaluronic acid, α-lipoic acid (ALA), magnesium, vitamin B6 and vitamin D, from the first visit at the experimental center (within the 12th week of gestation) for 3 months.
  Arms: Treatment group

SUMMARY:
The study aims to verify if the association of high molecular weight hyaluronic acid, α-lipoic acid (ALA), magnesium, vitamin B6 and vitamin D, reduces the risk of miscarriage in patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* two or more previous spontaneous first trimester abortions without apparent risk factors (idiopathic polyabortion)
* Endocrinopathies
* Autoimmune diseases
* Thrombophililic or coagulation diseases

Exclusion Criteria:

* Multiple pregnancies
* Presence of genetic abnormalities of one or both partners leading to increased risk of fetal aneuploidies
* Presence of Mullerian abnormalities in the uterus
* Symptoms present at recruitment such as pelvic pain or metrorrhagia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of metrorrhagia and/or pelvic pain in the first trimester of gestation. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Neuroscienze e Scienze riproduttive ed odontostomatologiche, Napoli, Italy